CLINICAL TRIAL: NCT07163455
Title: Time-Restricted Eating (10-Hour Window) for Weight-Loss Maintenance in Adults With Recent Intentional Weight Loss: A Multicenter, 12-Month Randomized Controlled Trial
Brief Title: Time-Restricted Eating for Weight-Loss Maintenance
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Harbin Medical University (Other)
Responsible Party: Principal Investigator, Ying Li, Professor, Harbin Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HMUIRB2025066PRE
Record Dates: First submitted 2025-08-14; First posted 2025-09-09 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Overweight or Obese Adults
MeSH Terms: conditions — Overweight

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Scheduled Weight Maintenance Nutrition Education (Active Comparator): Participants will receive standardized nutritional counseling for weight maintenance without any restriction on eating window. Dietary intake timing and body weight will be monitored using digital tracking tools throughout the study period.
  Interventions: Behavioral: Scheduled Weight Maintenance Nutrition Education
- Time-Restricted Eating (10-Hour Window) (Experimental): Same standardized sessions and monthly counseling as the control group, with the additional implementation of a 10-hour daily Time-Restricted Eating (TRE) regimen. Dietary intake timing and body weight will be monitored using digital tracking tools throughout the study period.
  Interventions: Behavioral: Time-Restricted Eating (10-Hour Window)

INTERVENTIONS:
Behavioral: Scheduled Weight Maintenance Nutrition Education — Participants will receive a standardized 30-45 minute weight maintenance nutrition education session at the time of randomization, covering principles of balanced dietary intake, reduction of salt, oil, and added sugar, adequate hydration. Thereafter, monthly 15-minute follow-up sessions will be delivered by trained dietitians, matched in frequency and content to those provided in the intervention arm. No temporal restriction will be imposed on eating behaviors. Participants will document meal intake via a mobile application using photograph-based entries with automated time-stamping and will record body weight weekly using Bluetooth-enabled digital scales. To ensure data accuracy, quality control will include twice-monthly brief telephone interviews for unannounced 24-hour dietary recalls.
  Arms: Scheduled Weight Maintenance Nutrition Education
Behavioral: Time-Restricted Eating (10-Hour Window) — In addition to receiving the same frequency and content of standardized nutritional counseling as the control group, participants will be instructed to confine all caloric intake to a self-selected 10-hour daily eating window. Outside of this window, only non-caloric beverages (e.g., water, unsweetened tea, black coffee) are permitted. Up to one exception day per week is allowed, during which intake may fall outside the designated window but must still be recorded. Dietary intake will be logged through a mobile application utilizing meal photographs with automated time-stamping; body weight will be recorded weekly using Bluetooth-enabled digital scales. As with the control group, participants will receive twice-monthly unannounced 24-hour dietary recalls and phone interviews to verify dietary records and ensure data quality.
  Arms: Time-Restricted Eating (10-Hour Window)

SUMMARY:
Weight regain after intentional short-term weight loss is a common challenge. It often undermines the long-term benefits of obesity treatment. This study is a multi-center 2-arm randomized controlled trial across six regions in China, specifically targeting overweight or obese adults who have recently achieved a short-term weight reduction (≥5% of body weight). The trial will evaluate whether a 10-hour daily Time-Restricted Eating (TRE) regimen can more effectively prevent weight regain compared to standard weight maintenance counseling alone. Both the intervention and control groups will receive the same frequency and intensity of nutritional counseling for weight maintenance; the only difference is that the TRE group will be instructed to confine their daily eating to a self-selected 10-hour window, while the control group has no eating window restriction. In addition to the primary outcome of weight regain, the study will explore potential mechanisms underlying the effects of TRE and assess secondary outcomes including changes in body composition, metabolic health, and quality of life.

This study recruits participants from six distinct regions across Eastern, Western, Southern, Northern, and Central China to enhance national representativeness. The study is divided into two phases: the first phase is a 2-month weight loss run-in phase (the screening phase), during which participants will receive standardized lifestyle and diet guidance from trained dietitians. Those who achieve at least a 5% loss of initial body weight by the end of this phase-and maintain a stable weight for approximately three weeks-will proceed to the second phase. In the second phase, participants will be randomly assigned to one of two arms for a 12-month weight maintenance intervention. The Control Arm will receive periodic weight-management nutritional counseling without any eating time restriction, while the TRE Intervention Arm will receive the same guidance plus instructions to follow a daily 10-hour time-restricted eating schedule. This design ensures both groups receive equivalent dietary and lifestyle support, with TRE as the key differential strategy. Following the 12-month intervention phase, participants will be followed for an additional 12 months (without active intervention) to observe longer-term weight outcomes.

Data will be collected at multiple time points: baseline (before the weight loss phase), 2 months (end of the weight loss phase and prior to the start of the maintenance phase), 5 months, 8 months, 14 months (end of the weight maintenance phase), as well as 20 months and 26 months (during the post-intervention follow-up). Key outcomes include changes in body weight (to assess weight regain or maintenance), body composition, metabolic health indicators (e.g. blood glucose, lipids), and quality of life measures. To monitor dietary behaviors, participants will be asked to upload meal photos via a designated mobile application with automatic time-stamping, which will be used to assess eating timing and adherence to the prescribed eating window. Body weight will be measured once weekly using Bluetooth-enabled smart scales. To explore potential mechanisms of action, biospecimens (blood and stool) will be collected at baseline, 2 months, 8 months, and 14 months for analysis. In addition, Continuous Glucose Monitoring (CGM) will be performed in a randomly selected subsample of 200 participants (100 from each group) using a standardized device for 14 consecutive days at months 2, 8, and 14. These data will be used to evaluate glycemic stability and adherence to the assigned eating window. Real-time CGM readings will not be disclosed to participants and will not be used to guide individual-level interventions.

ELIGIBILITY:
Inclusion Criteria:

* Participants who meet all the following conditions will be included in the trial:

  1. BMI ≥ 28.0 kg/m², or BMI between 24.0-27.9 kg/m² with at least one weight-related comorbidity.
  2. Age: 18-65 years.
  3. Weight Loss Plan: Willing to undergo a structured weight-loss program.

Exclusion Criteria:

* Participants who meet any of the following conditions will be excluded from the trial:

  1. Infectious Diseases: History of HIV/AIDS, active hepatitis B/C, or active tuberculosis.
  2. Malignancy: History of any malignancy.
  3. Organ Dysfunction:Severe hepatic impairment.Chronic kidney disease.
  4. Cardiovascular/Cerebrovascular Events: History of angina, myocardial infarction, or stroke within the past 6 months.
  5. Gastrointestinal Conditions:Severe gastrointestinal diseases (e.g., inflammatory bowel disease).Gastrointestinal surgery within the past 12 months.
  6. Endocrine Disorders:Cushing's syndrome, hypothyroidism, acromegaly, or hypothalamic obesity.
  7. Medications: Use of drugs affecting weight/energy balance (e.g., antipsychotics, weight-loss medications) within the past 6 months.
  8. Pregnancy/Lactation: Currently pregnant, planning pregnancy, or breastfeeding.
  9. Compliance Issues: Inability to complete the study (due to health, immigration, or other reasons).
  10. Informed Consent: Unwilling or unable to provide informed consent.
  11. Weight Stability: >5% change in body weight within the past 6 months.
  12. Individuals unable to use or operate a smartphone

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2026-01-26 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Weight change | At 0 (baseline), 2, 5, 8, 14, 20 and 26 months.
  The measurement will be conducted using the InBody570 bioelectrical impedance analyzer
Percentage of Participants Maintaining ≥5% Weight Loss from Baseline | At 14, 20, and 26 months
  The proportion of participants who achieve and sustain at least a 5% reduction in their baseline body weight by the end of the study. A participant is considered successful if their weight at 12 months is ≥5% lower than their weight at baseline.

SECONDARY OUTCOMES:
Change in waist circumference | At 0 (baseline), 2, 5, 8, 14, 20 and 26 months.
  Measurements will be taken using the same model of standardized soft measuring tape.
Change in hip circumference | At 0 (baseline), 2, 5, 8, 14, 20 and 26 months.
  Measurements will be taken using the same model of standardized soft measuring tape.
Change in body composition | At 0 (baseline), 2, 5, 8, 14, 20 and 26 months.
  The body composition of patients will be measured using the InBody570 bioelectrical impedance analyzer, assessing key parameters (e.g., body mass index [BMI], fat mass [FM], fat-free mass [FFM], skeletal muscle mass [SMM], visceral fat area [VFA], total body water [TBW], extracellular water [ECW], intracellular water [ICW], basal metabolic rate [BMR], waist-hip ratio [WHR], and phase angle [PhA]).
Change in blood pressure (systolic pressure and diastolic pressure) | At 0 (baseline), 2, 5, 8, 14, 20 and 26 months.
  Measurements will be taken using the same brand and model of precision blood pressure monitor.
Change in heart rate | At 0 (baseline), 2, 5, 8, 14, 20 and 26 months.
  Measurements will be taken using the same brand and model of precision blood pressure monitor.
Change in handgrip strength | At 0 (baseline), 2, 5, 8, 14, 20 and 26 months.
  The handgrip strength of patients will be assessed using handgrip dynamometers of the same brand and model.
Changes in blood transcriptomics | At 0 (baseline), 2, 8 and 14 months.
  Transcriptomic sequencing will be performed on blood samples collected from the patients to observe changes in blood transcriptional levels.
Changes in metabolomics in serum and feces | At 0 (baseline), 2, 8 and 14 months.
  Metabolomic sequencing will be performed on serum and fecal samples collected from the patients to observe changes in metabolic levels.
Change in quality of sleep measured by the Pittsburgh Sleep Quality Index (PSQI) | At 0 (baseline), 2, 5, 8, 14, 20 and 26 months.
  The sleep quality of each patient will be evaluated by the Pittsburgh Sleep Quality Index (PSQI), with scores ranging from 0 to 21, with higher scores indicating poorer sleep quality
Change in appetite states measured by the Electronic Visual Analogue Scale (eVAS) | At 0 (baseline), 2, 5, 8, 14, 20 and 26 months.
  Subjective appetite states were assessed using the Electronic Visual Analogue Scale (eVAS), with scores ranging from 0 to 100 for each dimension (hunger, fullness, desire to eat, and estimated food intake). Higher scores indicate stronger sensations.
The DISC Personality Assessment | At 0 (baseline)
  The DISC Personality Assessment evaluates four dimensions: Dominance (D), Influence (I), Steadiness (S), and Conscientiousness (C), with higher scores indicating stronger behavioral tendencies in each domain.
Change in quality of life measured by the Impact of Weight on Quality of Life-Lite (IWQOL-Lite) Questionnaire | At 0 (baseline), 2, 8, 14 and 26 months.
  Health-related quality of life was assessed using the Impact of Weight on Quality of Life-Lite (IWQOL-Lite) questionnaire, with scores ranging from 0 to 100 across five domains (Physical Function, Self-Esteem, Sexual Life, Public Distress, and Work Life). Higher scores indicate better weight-related quality of life.
Change in fasting blood glucose | At 0 (baseline), 2, 8 and 14 months.
  Blood samples from the patients will be tested for fasting blood glucose levels.
Change in fasting insulin | At 0 (baseline), 2, 8 and 14 months.
  Blood samples from the patients will be tested for fasting insulin levels.
Change in glycated hemoglobin (HbA1c) | At 0 (baseline), 2, 8 and 14 months.
  Blood samples from the patients will be tested for glycated hemoglobin (HbA1c) levels.
Change in serum creatinine level | At 0 (baseline), 2, 8 and 14 months.
  Serum creatinine level will be measured from blood samples using an enzymatic method. Results will be reported in micromoles per liter (μmol/L).
Change in blood urea nitrogen level | At 0 (baseline), 2, 8 and 14 months.
  Blood urea nitrogen level will be measured from blood samples using the urease method. Results will be reported in millimoles per liter (mmol/L).
Change in serum uric acid level | At 0 (baseline), 2, 8 and 14 months.
  Serum uric acid level will be measured from blood samples using the uricase-ultraviolet method. Results will be reported in micromoles per liter (μmol/L).
Change in serum Alanine Aminotransferase (ALT) level | At 0 (baseline), 2, 8 and 14 months.
  Serum alanine aminotransferase (ALT) level will be measured from blood samples using a rate method. Results will be reported in units per liter (U/L).
Change in serum Aspartate Aminotransferase (AST) level | At 0 (baseline), 2, 8 and 14 months.
  Serum aspartate aminotransferase (AST) level will be measured from blood samples using a rate method. Results will be reported in units per liter (U/L).
Change in Aspartate aminotransferase to Alanine aminotransferase ratio (AST/ALT) | At 0 (baseline), 2, 8 and 14 months.
  The AST/ALT ratio (De Ritis ratio) will be calculated from the measured values of serum aspartate aminotransferase (AST) and alanine aminotransferase (ALT). Results will be reported as a ratio.
Change in serum Gamma-Glutamyl Transferase (GGT) level | At 0 (baseline), 2, 8 and 14 months.
  Serum gamma-glutamyl transferase (GGT) level will be measured from blood samples using a rate method. Results will be reported in units per liter (U/L).
Change in serum Total Protein (TP) level | At 0 (baseline), 2, 8 and 14 months.
  Serum total protein (TP) level will be measured from blood samples using the biuret method. Results will be reported in grams per liter (g/L).
Change in serum Albumin (ALB) level | At 0 (baseline), 2, 8 and 14 months.
  Serum albumin (ALB) level will be measured from blood samples using the bromocresol green (BCG) method. Results will be reported in grams per liter (g/L).
Change in serum Globulin (GLOB) level | At 0 (baseline), 2, 8 and 14 months.
  Serum globulin (GLOB) level will be calculated by subtracting the measured serum albumin value from the measured serum total protein value. Results will be reported in grams per liter (g/L).
Change in Albumin to Globulin ratio (A/G) | At 0 (baseline), 2, 8 and 14 months.
  The Albumin to Globulin ratio (A/G) will be calculated from the measured values of serum albumin and calculated globulin. Results will be reported as a ratio.
Change in depression symptoms as measured by the Self-Rating Depression Scale (SDS) | At 0 (baseline), 2, 8, 14 and 26 months.
  Depression symptoms will be assessed using the Self-Rating Depression Scale (SDS). The SDS total score ranges from 20 to 80, with higher scores indicating more severe depressive symptoms (worse outcome).
Change in anxiety symptoms as measured by the Self-Rating Anxiety Scale (SAS) | At 0 (baseline), 2, 8, 14 and 26 months.
  Anxiety symptoms will be assessed using the Self-Rating Anxiety Scale (SAS). The SAS total score ranges from 20 to 80, with higher scores indicating more severe anxiety symptoms (worse outcome).
Change in serum Total Cholesterol (TC) level | At 0 (baseline), 2, 8 and 14 months.
  Serum concentration of Total Cholesterol (TC) will be measured from blood samples using the cholesterol oxidase method. Results will be reported in millimoles per liter (mmol/L).
Change in serum Triglycerides (TG) level | At 0 (baseline), 2, 8 and 14 months.
  Serum concentration of Triglycerides (TG) will be measured from blood samples using an enzymatic method. Results will be reported in millimoles per liter (mmol/L).
Change in serum High-Density Lipoprotein Cholesterol (HDL-C) level | At 0 (baseline), 2, 8 and 14 months.
  Serum concentration of High-Density Lipoprotein Cholesterol (HDL-C) will be measured from blood samples using an enzymatic method. Results will be reported in millimoles per liter (mmol/L).
Change in serum Low-Density Lipoprotein Cholesterol (LDL-C) level | At 0 (baseline), 2, 8 and 14 months.
  Serum concentration of Low-Density Lipoprotein Cholesterol (LDL-C) will be measured from blood samples using an enzymatic method. Results will be reported in millimoles per liter (mmol/L).
Change in serum Interleukin-1 beta (IL-1β) level | At 0 (baseline), 2, 8 and 14 months.
  Serum concentration of Interleukin-1 beta (IL-1β) will be measured from blood samples using a standardized multiplex immunoassay. Results will be reported in picograms per milliliter (pg/mL).
Change in serum Interleukin-6 (IL-6) level | At 0 (baseline), 2, 8 and 14 months.
  Serum concentration of Interleukin-6 (IL-6) will be measured from blood samples using a standardized multiplex immunoassay. Results will be reported in picograms per milliliter (pg/mL).
Change in serum Interleukin-8 (IL-8) level | At 0 (baseline), 2, 8 and 14 months.
  Serum concentration of Interleukin-8 (IL-8) will be measured from blood samples using a standardized multiplex immunoassay. Results will be reported in picograms per milliliter (pg/mL).
Change in serum Interleukin-10 (IL-10) level | At 0 (baseline), 2, 8 and 14 months.
  Serum concentration of Interleukin-10 (IL-10) will be measured from blood samples using a standardized multiplex immunoassay. Results will be reported in picograms per milliliter (pg/mL).
Change in serum Tumor Necrosis Factor-alpha (TNF-α) level | At 0 (baseline), 2, 8 and 14 months.
  Serum concentration of Tumor Necrosis Factor-alpha (TNF-α) will be measured from blood samples using a standardized multiplex immunoassay. Results will be reported in picograms per milliliter (pg/mL).
Change in serum Transforming Growth Factor-beta (TGF-β) level | At 0 (baseline), 2, 8 and 14 months.
  Serum concentration of Transforming Growth Factor-beta (TGF-β) will be measured from blood samples using a standardized multiplex immunoassay. Results will be reported in picograms per milliliter (pg/mL).
Change in serum Monocyte Chemoattractant Protein-1 (MCP-1/CCL2) level | At 0 (baseline), 2, 8 and 14 months.
  Serum concentration of Monocyte Chemoattractant Protein-1 (MCP-1/CCL2) will be measured from blood samples using a standardized multiplex immunoassay. Results will be reported in picograms per milliliter (pg/mL).
Change in serum Leptin level | At 0 (baseline), 2, 8 and 14 months.
  Serum concentration of Leptin will be measured from blood samples using a standardized immunoassay. Results will be reported in nanograms per milliliter (ng/mL).
Change in serum Adiponectin level | At 0 (baseline), 2, 8 and 14 months.
  Serum concentration of Adiponectin will be measured from blood samples using a standardized immunoassay. Results will be reported in micrograms per milliliter (μg/mL).
Change in serum C-reactive Protein (CRP) level | At 0 (baseline), 2, 8 and 14 months.
  Serum concentration of C-reactive Protein (CRP) will be measured from blood samples using an immunoturbidimetric assay. Results will be reported in milligrams per liter (mg/L).
Change in serum Tumor Necrosis Factor-alpha-induced protein 3 (TNFAIP3/A20) level | At 0 (baseline), 2, 8 and 14 months.
  Serum concentration of Tumor Necrosis Factor-alpha-induced protein 3 (TNFAIP3/A20) will be measured from blood samples using a standardized enzyme-linked immunosorbent assay (ELISA). Results will be reported in nanograms per milliliter (ng/mL).
Change in plasma Lipopolysaccharide (LPS) level | At 0 (baseline), 2, 8 and 14 months.
  Plasma concentration of Lipopolysaccharide (LPS) will be measured from blood samples using a commercial enzyme-linked immunosorbent assay (ELISA) kit. Results will be reported in endotoxin units per milliliter (EU/mL).
Change in serum Lipopolysaccharide-Binding Protein (LBP) level | At 0 (baseline), 2, 8 and 14 months.
  Serum concentration of Lipopolysaccharide-Binding Protein (LBP) will be measured from blood samples using a commercial enzyme-linked immunosorbent assay (ELISA) kit. Results will be reported in micrograms per milliliter (μg/mL).
Change in serum Resolvin D1 (RvD1) level | At 0 (baseline), 2, 8 and 14 months.
  Serum concentration of Resolvin D1 (RvD1) will be measured from blood samples using liquid chromatography with tandem mass spectrometry (LC-MS/MS). Results will be reported in picograms per milliliter (pg/mL).
Change in serum Resolvin E1 (RvE1) level | At 0 (baseline), 2, 8 and 14 months.
  Serum concentration of Resolvin E1 (RvE1) will be measured from blood samples using liquid chromatography with tandem mass spectrometry (LC-MS/MS). Results will be reported in picograms per milliliter (pg/mL).
Daily Energy and Macronutrient Intake | At 0 (baseline), 2, 5, 8 14, 20, and 26 months.
  Total energy intake and macronutrient distribution (percentage of energy from carbohydrates, fat, and protein) will be assessed at each time point using three non-consecutive 24-hour dietary recalls. Results will be reported in kilocalories (kcal) for energy and percentage points (%) for macronutrient distribution.
Within-individual variability in daily interstitial glucose (SD) | At months 2, 8, and 14. Each assessment will be conducted using continuous glucose monitoring (CGM) over a consecutive 14-day period.
  Variability in daily interstitial glucose will be assessed using the standard deviation (SD) of mean daily glucose values across the continuous glucose monitoring (CGM) period. This metric quantifies day-to-day fluctuation in glucose concentration. Results will be reported in milligrams per deciliter (mg/dL).
Within-individual variability in daily interstitial glucose (CV) | At months 2, 8, and 14. Each assessment will be conducted using continuous glucose monitoring (CGM) over a consecutive 14-day period.
  Variability in daily interstitial glucose will be assessed using the coefficient of variation (CV), calculated as the standard deviation divided by the mean glucose level across the CGM period. This metric quantifies relative variability in glucose concentration. Results will be reported as a percentage (%).
Mean amplitude of glycemic excursions (MAGE) | At months 2, 8, and 14. Each assessment will be conducted using continuous glucose monitoring (CGM) over a consecutive 14-day period.
  Variability in daily interstitial glucose will be assessed using mean amplitude of glycemic excursions (MAGE), which represents the average magnitude of significant glucose fluctuations across the CGM period. This metric quantifies short-term glycemic variability. Results will be reported in milligrams per deciliter (mg/dL).
Percentage of monitoring time with interstitial glucose 70-140 mg/dL (TIR) | At months 2, 8, and 14. Each assessment will be conducted using continuous glucose monitoring (CGM) over a consecutive 14-day period.
  Glycemic control will be assessed as the percentage of total monitoring time spent in the target glucose range of 70-140 mg/dL during CGM. This metric quantifies the proportion of time glucose values remain within the predefined range. Results will be reported as a percentage (%).
Change in postprandial glucose excursion | At 2, 8, and 14 months.
  The magnitude of postprandial glucose excursion will be assessed using continuous glucose monitoring (CGM), calculated as the difference between the peak interstitial glucose concentration and the pre-prandial level following main meals. Glucose data will be time-synchronized with self-reported dietary intake logs. Results will be reported in millimoles per liter (mmol/L).
Change in postprandial time above range (pTAR) | At 2, 8, and 14 months.
  The percentage of time that interstitial glucose concentrations exceed 10.0 mmol/L during the 3-hour postprandial period will be assessed using continuous glucose monitoring (CGM). Glucose data will be time-synchronized with self-reported dietary intake logs. Results will be reported as a percentage of the postprandial monitoring period (%).
Change in thyroid-stimulating hormone (TSH) | At 0 (baseline), 2, 8 and 14 months.
  Serum TSH levels will be measured from blood samples. Results will be reported in milli-international units per liter (mIU/L).
Change in free thyroxine (FT4) | At 0 (baseline), 2, 8 and 14 months.
  Serum FT4 levels will be measured from blood samples. Results will be reported in picomoles per liter (pmol/L).
DNA Methylation Patterns | At 0 (baseline), 2, 8, and 14 months.
  Genome-wide DNA methylation profiles will be assessed using peripheral blood samples collected at specified time points. Changes in DNA methylation will be explored as potential mechanistic biomarkers mediating the effects of time-restricted eating on metabolic health and weight regulation.

CONTACTS AND LOCATIONS:
Locations (10):
- China (10):
  - Shenzhen People's Hospital, Shenzhen, Guangdong
  - Peking University Shenzhen Hospital, Shenzhen, Guangdong
  - The First Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Harbin Medical University, Harbin, Heilongjiang
  - The Second Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - The Second Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Weifang People's Hospital, Weifang, Shandong
  - Air Force Hospital of Western Theater Command,PLA, Chengdu, Sichuan
  - Chengdu Seventh People's Hospital, Chengdu, Sichuan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jakubowicz D, Barnea M, Wainstein J, Froy O. High caloric intake at breakfast vs. dinner differentially influences weight loss of overweight and obese women. Obesity (Silver Spring). 2013 Dec;21(12):2504-12. doi: 10.1002/oby.20460. Epub 2013 Jul 2. PMID 23512957
- [Background] Mentzelou M, Papadopoulou SK, Psara E, Voulgaridou G, Pavlidou E, Androutsos O, Giaginis C. Chrononutrition in the Prevention and Management of Metabolic Disorders: A Literature Review. Nutrients. 2024 Mar 1;16(5):722. doi: 10.3390/nu16050722. PMID 38474850
- [Background] Wilkinson MJ, Manoogian ENC, Zadourian A, Lo H, Fakhouri S, Shoghi A, Wang X, Fleischer JG, Navlakha S, Panda S, Taub PR. Ten-Hour Time-Restricted Eating Reduces Weight, Blood Pressure, and Atherogenic Lipids in Patients with Metabolic Syndrome. Cell Metab. 2020 Jan 7;31(1):92-104.e5. doi: 10.1016/j.cmet.2019.11.004. Epub 2019 Dec 5. PMID 31813824
- [Background] Reytor-Gonzalez C, Simancas-Racines D, Roman-Galeano NM, Annunziata G, Galasso M, Zambrano-Villacres R, Verde L, Muscogiuri G, Frias-Toral E, Barrea L. Chrononutrition and Energy Balance: How Meal Timing and Circadian Rhythms Shape Weight Regulation and Metabolic Health. Nutrients. 2025 Jun 27;17(13):2135. doi: 10.3390/nu17132135. PMID 40647240
- [Background] Liu HY, Eso AA, Cook N, O'Neill HM, Albarqouni L. Meal Timing and Anthropometric and Metabolic Outcomes: A Systematic Review and Meta-Analysis. JAMA Netw Open. 2024 Nov 4;7(11):e2442163. doi: 10.1001/jamanetworkopen.2024.42163. PMID 39485353
- [Background] Duez H, Staels B. Circadian Disruption and the Risk of Developing Obesity. Curr Obes Rep. 2025 Feb 13;14(1):20. doi: 10.1007/s13679-025-00610-6. PMID 39939483
- [Background] Ruddick-Collins LC, Morgan PJ, Fyfe CL, Filipe JAN, Horgan GW, Westerterp KR, Johnston JD, Johnstone AM. Timing of daily calorie loading affects appetite and hunger responses without changes in energy metabolism in healthy subjects with obesity. Cell Metab. 2022 Oct 4;34(10):1472-1485.e6. doi: 10.1016/j.cmet.2022.08.001. Epub 2022 Sep 9. PMID 36087576
- [Background] Thomas JG, Panza E, Goldstein CM, Hayes JF, Benedict N, O'Leary K, Wing RR. Pragmatic Implementation of Online Obesity Treatment and Maintenance Interventions in Primary Care: A Randomized Clinical Trial. JAMA Intern Med. 2024 May 1;184(5):502-509. doi: 10.1001/jamainternmed.2023.8438. PMID 38466266
- [Background] Gill S, Le HD, Melkani GC, Panda S. Time-restricted feeding attenuates age-related cardiac decline in Drosophila. Science. 2015 Mar 13;347(6227):1265-9. doi: 10.1126/science.1256682. PMID 25766238
- [Background] Apolzan JW, Venditti EM, Edelstein SL, Knowler WC, Dabelea D, Boyko EJ, Pi-Sunyer X, Kalyani RR, Franks PW, Srikanthan P, Gadde KM; Diabetes Prevention Program Research Group. Long-Term Weight Loss With Metformin or Lifestyle Intervention in the Diabetes Prevention Program Outcomes Study. Ann Intern Med. 2019 May 21;170(10):682-690. doi: 10.7326/M18-1605. Epub 2019 Apr 23. PMID 31009939
- [Background] Kim JY. Optimal Diet Strategies for Weight Loss and Weight Loss Maintenance. J Obes Metab Syndr. 2021 Mar 30;30(1):20-31. doi: 10.7570/jomes20065. PMID 33107442
- [Background] Ludwig DS, Ebbeling CB. Weight-loss maintenance--mind over matter? N Engl J Med. 2010 Nov 25;363(22):2159-61. doi: 10.1056/NEJMe1011361. No abstract available. PMID 21105799
- [Background] Sacks FM, Bray GA, Carey VJ, Smith SR, Ryan DH, Anton SD, McManus K, Champagne CM, Bishop LM, Laranjo N, Leboff MS, Rood JC, de Jonge L, Greenway FL, Loria CM, Obarzanek E, Williamson DA. Comparison of weight-loss diets with different compositions of fat, protein, and carbohydrates. N Engl J Med. 2009 Feb 26;360(9):859-73. doi: 10.1056/NEJMoa0804748. PMID 19246357
- [Background] Kadam I, Neupane S, Wei J, Fullington LA, Li T, An R, Zhao L, Ellithorpe A, Jiang X, Wang L. A Systematic Review of Diet Quality Index and Obesity among Chinese Adults. Nutrients. 2021 Oct 11;13(10):3555. doi: 10.3390/nu13103555. PMID 34684556
- [Background] Wang L, Zhou B, Zhao Z, Yang L, Zhang M, Jiang Y, Li Y, Zhou M, Wang L, Huang Z, Zhang X, Zhao L, Yu D, Li C, Ezzati M, Chen Z, Wu J, Ding G, Li X. Body-mass index and obesity in urban and rural China: findings from consecutive nationally representative surveys during 2004-18. Lancet. 2021 Jul 3;398(10294):53-63. doi: 10.1016/S0140-6736(21)00798-4. PMID 34217401
- [Background] Sun Z, Sun M, Wei W, Peng W, Wang Y. China launches National Obesity Campaign. Lancet Diabetes Endocrinol. 2025 Jun;13(6):465-466. doi: 10.1016/S2213-8587(25)00131-7. No abstract available. PMID 40404276